CLINICAL TRIAL: NCT06120673
Title: International, Multi-centre Randomised Clinical Trial of Obinutuzumab Versus Corticosteroid and Cyclophosphamide in Primary Membranous Nephropathy (REMIT Trial).
Brief Title: REmission in Membranous Nephropathy International Trial (REMIT)
Acronym: REMIT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was deemed unfeasible due to unforeseen financial limitations
Sponsor: The University of Queensland (Other)
Collaborators: University of Adelaide (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKTN 18.03
Record Dates: First submitted 2022-12-12; First posted 2023-11-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-04

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — obinutuzumab; Prednisolone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obinutuzumab (Experimental)
  Interventions: Drug: Obinutuzumab
- Oral prednisolone and cyclophosphamide (Active Comparator)
  Interventions: Drug: Oral prednisolone and cyclophosphamide

INTERVENTIONS:
Drug: Obinutuzumab — Participants will receive an intravenous infusion of 1,000mg Obinutuzumab at Weeks 0, 2, 24 and 26.
  Prior to the administration of obinutuzumab, the participant will receive pre-medications consisting of all three:
  * IV methylprednisolone 80 mg,
  * Paracetamol 1,000 mg orally,
  * Either cetirizine 10 mg orally or diphenhydramine 50 mg orally. These pre-medications must be completed between 30 to 60 minutes prior to the obinutuzumab infusion.
  Arms: Obinutuzumab
Drug: Oral prednisolone and cyclophosphamide — Participants will receive a combination of oral prednisolone and cyclophosphamide with 2 options (Option A and B).
  Option A: Cyclical prednisolone and cyclophosphamide with IV methylprednisolone
  * IV methylprednisolone 500-1000 mg will be given on days 1, 2 and 3 at the start of months 1, 3, and 5.
  * Oral prednisolone will be given at 0.5 mg/kg/day (max 50 mg/day) in months 1, 3, and 5.
  * Oral cyclophosphamide will be given in months 2, 4 and 6, adjusted by age and weight
  Option B: Concurrent prednisolone and cyclophosphamide without IV methylprednisolone
  * Oral prednisolone will be given to meet a cumulative dose equivalent to 0.5 mg/kg/day for 90 days (max 50 mg/day).
  * Oral cyclophosphamide will be given for 90 days, adjusted by age and weight
  Arms: Oral prednisolone and cyclophosphamide

SUMMARY:
REMIT is an investigator-initiated, international, multi-centre, prospective, randomised, open-label, parallel-group trial. A total of 224 adult participants with Primary Membranous Nephropathy (PMN) will be recruited from renal units from Australia, New Zealand Canada, Asia, Europe, United Kingdom, and other countries. Participants will be randomised to receive either corticosteroid and cyclophosphamide or obinutuzumab. The primary outcome is a ranked, composite measure based on (a) efficacy, defined as either complete or partial remission of PMN, (b) number of adverse events, and (c) quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Able to provide informed consent.
3. Primary Membranous Nephropathy (PMN) confirmed by:

   1. Kidney biopsy (anti-PLA2R negative patients are eligible for inclusion if PMN is confirmed on biopsy. Kidney biopsy is generally encouraged to confirm diagnosis of PMN) or
   2. if the clinician decides against a biopsy, the patient must be anti-PLA2R positive and must not have diabetes.
4. Proteinuria ≥4 g/24h despite supportive treatment for at least 6 months with maximally tolerated dose of ACE-i or ARB (dose to be stable for at least 4 weeks), confirmed at final screening before randomisation
5. Serum albumin <30 g/L.
6. Estimated glomerular filtration rate (eGFR) ≥40 ml/min/1.73m2.
7. Treatment with immunosuppression is warranted, as determined by the treating physician.
8. Fully vaccinated against COVID-19 according to local practice/recommendation.

Exclusion Criteria:

1. Resistant to rituximab or have had >2 g of rituximab in the past.
2. Resistant to cyclophosphamide or have had a cumulative >20 g of cyclophosphamide in the past.
3. More than 3 years since PMN diagnosis.
4. Proteinuria must not have decreased by >50% over 6 months whilst taking ACE-i/ARB.
5. Patients with human immunodeficiency virus (HIV) infection, active hepatitis B or C infection, or other active infections.
6. Patients with secondary membranous nephropathy
7. Screening for malignancy must be considered especially in cases who are anti-PLA2R negative.
8. Patients whose kidney biopsy shows concomitant features of diabetic nephropathy.
9. Kidney transplant recipients.
10. Pregnancy or breastfeeding.
11. Women of childbearing age not willing to use contraception.
12. Suspected or known hypersensitivity, allergy, and/or immunogenic reaction history to monoclonal antibodies, corticosteroid, cyclophosphamide, any of their ingredients, and any other drugs from these same pharmacotherapeutic groups.
13. Any disorder or condition, in the opinion of the investigator, might pose an unacceptable risk to participant's safety and well-being.
14. Inability to understand or comply with the requirements of the study.
15. Incapable of recognizing the nature, significance, and scope of the clinical trial or giving consent are excluded, even if they have a legal representative.
16. Use of an investigational agent <30 days or within five half-lives of the investigational agents (whichever is longer), whose effect or toxicity may overlap with that of obinutuzumab, prednisolone, cyclophosphamide, or their metabolites.
17. Active Tuberculosis infection. Testing for latent disease may be performed at screening if required by local regulations or in accordance with local clinical practice. Latent disease after completion of appropriate treatment is not exclusionary.
18. Low peripheral B-cell count (as per local reference range) . B-cell count must be checked, particularly in those who have received rituximab, cyclophosphamide or both anytime in the past.
19. Use of SGLT2-i and GLP-1 agonist within 90 days prior to randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
A ranked composite measure based efficacy, safety and quality of life at 24 months | 24 months
  A ranked composite measure comprising of:
  1. Efficacy (complete/partial remission) plus safety (type of adverse event) at 24 months
  2. Number of adverse events up to 24 months
  3. Quality of Life (EQ-5D) averaged over 24 months

SECONDARY OUTCOMES:
Number of participants in Complete Remission (CR) | At 6, 12, 18, 24 month
  Number of participants who have proteinuria of ≤3.0 g/day
Number of participants in Partial Remission (PR) | At 6, 12, 18, 24 month
  Number of participants who have proteinuria of between >3.0 and 3.5 g/day and >50% reduction from baseline proteinuria
Number of participants in CR and/or PR | At 6, 12, 18, 24 month
  Number of participants who meet complete and/or partial PMN remission definition
Number of non-serious adverse events of special interest | Up until 24 months
  Number of protocol defined non-serious events of special interest (related to PMN or the study interventions)
Number of serious adverse events | Up until 24 months
  Number of protocol defined serious adverse events
Number of participants with a lack of response to PMN treatment | Up until 24 months
  Number of participants who have <50% reduction in proteinuria from baseline or worsening (increasing in value from baseline) proteinuria, and had not achieved either PR or CR
Number of participants who relapse after CR or PR | Up until 24 months
  Number of participant who have a reappearance of proteinuria to >3.5 g/day at a ≥50% higher level than the lowest post-treatment value in participants who had previously achieved either PR or CR
Time to first relapse | Up until 24 months
  The time to relapse is the time interval from the last point in time when the participant was in the best remission status (either PR or CR) to the first relapse
Number of participants who have immunological remission (for anti-PLA2R positive participants) | Up until 24 months
  Number of participants who have their anti-PLA2R-Ab level drop below 2 RU/mL who are ≥14 RU/ml at baseline
Number of participants who have a requirement for rescue therapy | Up until 24 months
  Number of participants who have a lack of response or relapse at 12 months, and rescue therapies such as obinutuzumab, calcineurin inhibitors, or additional corticosteroid and cyclophosphamide are used.
Number of participants who exit the trial | Up until 24 months
  Number participant who cease trial follow-up for any reason
Quality of life scores (EQ-5D-5L) | at 3, 6, 9, 12, 15, 18, 24 months
  Quality of life scores using EQ-5D-5L
eGRF slope | Up until 24 months
  Change in eGFR slope
Number of treatment or PMN associated deaths | Up until 24 months
  Number of deaths attributed directly or indirectly to a complication of PMN or the treatment for PMN
All cause deaths | Up until 24 months
  Number of deaths of any cause

OTHER OUTCOMES:
Number of participants in Complete Remission (CR) | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Number of participants who have proteinuria of ≤3.0 g/day
Number of participants in Partial Remission (PR) | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Number of participants who have proteinuria of between >3.0 and 3.5 g/day and >50% reduction from baseline proteinuria with stable kidney function (eGFR remains >40 ml/min/1.73m2)
Number of participants in CR and/or PR | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Number of participants who meet complete and/or partial PMN remission definition
Number of non-serious adverse events of special interest | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Number of protocol defined non-serious events of special interest (related to PMN or the study interventions)
Number of serious adverse events | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Number of protocol defined serious adverse events
Number of participants with a lack of response to PMN treatment | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Number of participants who have <50% reduction in proteinuria from baseline or worsening (increasing in value from baseline) proteinuria, and had not achieved either PR or CR
Number of participants who have immunological remission (for anti-PLA2R positive participants) | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Number of participants who have their anti-PLA2R-Ab level drop below 2 RU/mL who are ≥14 RU/ml at baseline
Requirement for dialysis or kidney transplant | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Number of participants who require dialysis or a kidney transplant (Stage 5 kidney disease)
eGRF slope | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Change in eGFR slope
Number of participants with treatment or PMN associated death | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Number of deaths attributed directly or indirectly to a complication of PMN or the treatment for PMN
Number of participants with all cause death | At any point up until end of study (when last participant reaches 24 months - ~42 months)
  Number of deaths of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Chen Au Peh, Study Chair — The University of Adelaide; Bhadran Bose, Study Director — Nepean Blue Mountains Local Health District
Locations (13):
- Australia (13):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Bundaberg Hospital, Bundaberg, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Logan Hospital, Logan City, Queensland
  - Mackay Base Hospital, Mackay, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - Mater Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Fiona Stanley Hospital, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Data sets will be made available to researchers within the REMIT Study for analysis of sub-studies and country specific outcomes after the primary manuscript has been accepted for publication.
  For researchers outside the REMIT study, individual participant data will be made available upon request to a Data Access Committee, a review board set up to assess proposals based on sound science, benefit-risk balancing and research team expertise.
  Where data linkage has been used to estimate health care services utilisation, data sharing will be determined by the specific requirements of the data custodians. In some circumstances it may not be possible to share participant level data beyond the country in which it was collected. This will be addressed on a jurisdiction basis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after publication of pre-specified analyses
Access Criteria: Data sets will be made available to researchers within the REMIT Study for analysis of sub-studies and country specific outcomes after the primary manuscript has been accepted for publication.
  For researchers outside the REMIT study, individual participant data will be made available upon request to a Data Access Committee, a review board set up to assess proposals based on sound science, benefit-risk balancing and research team expertise.